CLINICAL TRIAL: NCT06332352
Title: Intra-articular Platelet-Rich Plasma in the Management of Acetabular Labral Tears: a Prospective Study
Brief Title: Intra-articular Platelet-Rich Plasma for Acetabular Labral Tears
Acronym: PRP for ALT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00173470
Record Dates: First submitted 2024-03-01; First posted 2024-03-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Acetabular Labrum Tear
Keywords: Acetabular Labrum Tear; Platelet Rich Plasma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-Articular hip injection of PRP (Experimental): Single Group Assignment Recruitment will occur at the University of Utah Orthopedic Center by physician and study staff members medical chart review before patient visits. 45 mL of blood will be collected from eligible participants and processed. A single processed neutrophil-poor PRP injection will be given once to a single hip.
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — Intra-articular hip injection of PRP, Blood Collection 45mL, Processed Neutrophil-Poor PRP, 1 injection to one hip joint.

SUMMARY:
Platelets are small cells found in the blood that help form clots and stop bleeding. Platelet-rich plasma is blood that contains more platelets than normal and can be given to help people with pain. Tears of the Labrum to the hip (the cartilage "suction cup" that holds the ball to the socket of the hip) cause hip pain. The study wants to see if a portion of the patient's blood, the platelets, will help relieve hip pain and function.

Participation requires completing surveys by email, text message, in person, and/or by telephone. Medical tests will also be done to track the health of participants.

DETAILED DESCRIPTION:
Acetabular labral tears (ALT) have been reported to have a prevalence of 22-55% in patients presenting with hip or groin pain. Etiologies of ALT include femoral acetabular impingement (FAI) as the most common followed by trauma, degeneration, dysplasia, hypermobility, etc. The fibrocartilaginous acetabular labrum is an important structure in the maintenance of hip perseveration and biomechanics. Several functions include decreasing stress on articular surfaces by increasing surface contact area, maintaining a pressurized layer of intra-articular fluid to distribute mechanical forces, and assisting in joint stability. The consequences of labral pathology are not fully understood, however, prior studies have indicated that there is a correlation between acetabular labral lesions and chondral injury contributing to the development of early degenerative hip disease.

Based on current evidence, it is suggested that the highest degree of clinical accuracy in the diagnosis of a symptomatic acetabular labral tear is with a combination of clinical history, physical examination, advanced imaging such as magnetic resonance imaging (MRI) or magnetic resonance angiography (MRA), and diagnostic injection. Conservative management trials are often considered for initial treatment and include relative rest, activity modification, anti-inflammatory medication, and physical therapy with the potential for intra-articular injections including corticosteroids. If conservative management is unsuccessful, arthroscopic intervention with resection, refixation, or reconstruction is often considered. If conservative management is unsuccessful, arthroscopic intervention with resection, refixation, or reconstruction is often considered.

According to a recent systematic review and meta-analysis, there is promising evidence that platelet rich plasma (PRP) is an effective treatment for hip osteoarthritis. However, there is limited evidence regarding PRP treatment for ALT. To date, there is only one pilot study published evaluating 8 patients diagnosed with ALT who underwent ultrasound guided intra-articular hip injection with PRP. Optimistically, this study did reveal significant differences from baseline in function and pain scores at short term follow-up. However, the study lacked many important details including information about the injectate (the composition of the blood and PRP) which is vital to include in studies of these types. Therefore, the purpose of this study is to fully evaluate the effects of PRP treatment on the clinical outcomes of ALT prospectively in a larger cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤49 years old (i.e., 18 - 49 years old)
* Hip or groin pain with at least 1 positive provocative labral hip maneuver (i.e., Flexion, Adduction, Internal Rotation (FADIR) test, subspine impingement test, scour)
* Radiographs with Tonnis grade < 2 (i.e., 0 or 1)
* MRI or MRA hip with evidence of acetabular labral tear
* Failure of at least 6 weeks of conservative management [i.e., activity modification, non-steroidal anti-inflammatory drugs (NSAIDs), and/or physical therapy (PT), other intra-articular injection etc.]
* Prior diagnostic ultrasound guided hip injection with anesthetic-only providing ≥50% pain relief

Exclusion Criteria:

* Any prior surgery to the affected hip
* Imaging with evidence of avascular necrosis of the affected hip
* Imaging with evidence of hip dysplasia (i.e. lateral center edge angle of ≤20 degrees)
* Alpha angle of ≥55 degrees of the affected hip
* Intra-articular hip injection within the last 6 months to the affected hip of any injectate with the exception of anesthetic
* Active systemic infection requiring antibiotics or local infection at the site of the injection
* Any prior intra-articular infection of the affected hip
* Any prior fracture of the affected femur or pelvis
* Blood dyscrasia or malignancy
* Non-ambulatory patients
* Patient seeking care with active litigation pending
* Body mass index (BMI) ≥ 35 kg/m2
* Systemic inflammatory arthropathy
* Oral steroids consumed within the last three months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Pain & Function Improvements | 12 Months
  The primary analysis will be an improvement in Harris Hip Scores (HHS) and Visual Analog Scale (VAS) over twelve months. Descriptive statistics will be calculated for patent demographics and clinical characteristics as well as for pre-injection (baseline) and post-injection (at 1, 3, 6, and 12 months) data for VAS and HHS.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  VAS at 1, 3, 6, and 12 months after injection. The VAS asks "Overall, how would you rate your hip from 0 (worst possible) - 100 (best possible)".
Harris Hip Scores (HHS) | 12 Months
  Harris Hip Scores (HHS) at 1,3, 6, and 12 months after their injection. There are ten items covering four domains. The domains are pain, function, absence of deformity, and range of motion.
  The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
International Hip Outcome Tool (iHOT-12) | 12 Months
  International Hip Outcome Tool (iHOT-12) at 1, 3, 6, and 12 months after their injection. The iHOT-12 consists of four domains; symptoms and functional limitations, sport and recreational activities, job-related concerns, and social, emotional, and lifestyle concerns.
  Each item in the iHOT-12 was scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms, and the overall mean equates to the final iHOT score.
EQ-5D (EuroQual 5D) | 12 Months
  EQ-5D (EuroQual 5D) at 1, 3, 6, and 12 months after their injection. The EQ-5D consists of 5 domains; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each of the 5 domains are divided into 5 levels of problems (Level 1: indicating no problems, Level 2: indicating slight problems, Level 3: indicating moderate problems, Level 4: indicating severe problems, and Level 5: indicating extreme problems). The EQ-5D also includes an overall health domain rated from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cushman, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah - Department of Orthopaedics, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Groh MM, Herrera J. A comprehensive review of hip labral tears. Curr Rev Musculoskelet Med. 2009 Jun;2(2):105-17. doi: 10.1007/s12178-009-9052-9. Epub 2009 Apr 7. PMID 19468871
- [Background] Ishoi L, Nielsen MF, Krommes K, Husted RS, Holmich P, Pedersen LL, Thorborg K. Femoroacetabular impingement syndrome and labral injuries: grading the evidence on diagnosis and non-operative treatment-a statement paper commissioned by the Danish Society of Sports Physical Therapy (DSSF). Br J Sports Med. 2021 Nov;55(22):1301-1310. doi: 10.1136/bjsports-2021-104060. Epub 2021 Sep 16. PMID 34531185
- [Background] Bsat S, Frei H, Beaule PE. The acetabular labrum: a review of its function. Bone Joint J. 2016 Jun;98-B(6):730-5. doi: 10.1302/0301-620X.98B6.37099. PMID 27235512
- [Background] Su T, Chen GX, Yang L. Diagnosis and treatment of labral tear. Chin Med J (Engl). 2019 Jan 20;132(2):211-219. doi: 10.1097/CM9.0000000000000020. PMID 30614856
- [Background] McCarthy JC, Noble PC, Schuck MR, Wright J, Lee J. The Otto E. Aufranc Award: The role of labral lesions to development of early degenerative hip disease. Clin Orthop Relat Res. 2001 Dec;(393):25-37. doi: 10.1097/00003086-200112000-00004. PMID 11764355
- [Background] Chinzei N, Hashimoto S, Hayashi S, Takayama K, Matsumoto T, Kuroda R. Prediction of intra-articular pathology and arthroscopic outcomes for femoroacetabular impingement and labral tear based on the response to preoperative anaesthetic hip joint injections. Eur J Orthop Surg Traumatol. 2020 May;30(4):737-742. doi: 10.1007/s00590-020-02627-0. Epub 2020 Jan 20. PMID 31960159
- [Background] Yoong P, Guirguis R, Darrah R, Wijeratna M, Porteous MJ. Evaluation of ultrasound-guided diagnostic local anaesthetic hip joint injection for osteoarthritis. Skeletal Radiol. 2012 Aug;41(8):981-5. doi: 10.1007/s00256-011-1290-4. Epub 2011 Nov 10. PMID 22069031
- [Background] Byrd JW, Jones KS. Diagnostic accuracy of clinical assessment, magnetic resonance imaging, magnetic resonance arthrography, and intra-articular injection in hip arthroscopy patients. Am J Sports Med. 2004 Oct-Nov;32(7):1668-74. doi: 10.1177/0363546504266480. PMID 15494331
- [Background] O'Dowd A. Update on the Use of Platelet-Rich Plasma Injections in the Management of Musculoskeletal Injuries: A Systematic Review of Studies From 2014 to 2021. Orthop J Sports Med. 2022 Dec 9;10(12):23259671221140888. doi: 10.1177/23259671221140888. eCollection 2022 Dec. PMID 36532150
- [Background] Saied AM, Redant C, El-Batouty M, El-Lakkany MR, El-Adl WA, Anthonissen J, Verdonk R, Audenaert EA. Accuracy of magnetic resonance studies in the detection of chondral and labral lesions in femoroacetabular impingement: systematic review and meta-analysis. BMC Musculoskelet Disord. 2017 Feb 16;18(1):83. doi: 10.1186/s12891-017-1443-2. PMID 28209142
- [Background] Conaway Wea. Predictors of Outcomes of Non-Surgical Management for Acetabular Labral Tears. Orthopaedic Journal of Sports Medicine. 2018;6(3).
- [Background] Lim A, Zhu JB, Khanduja V. The Use of Intra-articular Platelet-Rich Plasma as a Therapeutic Intervention for Hip Osteoarthritis: A Systematic Review and Meta-analysis. Am J Sports Med. 2023 Jul;51(9):2487-2497. doi: 10.1177/03635465221095563. Epub 2022 Jun 7. PMID 35971803
- [Background] De Luigi AJ, Blatz D, Karam C, Gustin Z, Gordon AH. Use of Platelet-Rich Plasma for the Treatment of Acetabular Labral Tear of the Hip: A Pilot Study. Am J Phys Med Rehabil. 2019 Nov;98(11):1010-1017. doi: 10.1097/PHM.0000000000001237. PMID 31162277